CLINICAL TRIAL: NCT03915379
Title: A Phase 1, First-in-Human, Open-Label, Dose Escalation Study of JNJ-67371244 (Bispecific Antibody Targeting CD33 and CD3), in Subjects With Relapsed or Refractory Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS)
Brief Title: A Study of JNJ-67571244 in Participants With Relapsed or Refractory Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108582; 2018-004452-37 (EudraCT Number); 67571244AML1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-03-29; First posted 2019-04-16 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Leukemia, Myeloid, Acute; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): Participants will receive JNJ-67571244. The dose levels will be escalated sequentially based on the decisions of the Study Evaluation Team (SET) until the recommended Phase 2 Dose (RP2D) has been identified.
  Interventions: Drug: JNJ-67571244
- Part 2: Dose Expansion (Experimental): Participants in 2 expansion cohorts of acute myeloid leukemia (AML) or either high-risk myelodysplastic syndromes (MDS) or very high-risk MDS will receive JNJ-67571244 at the RP2D determined in Part 1.
  Interventions: Drug: JNJ-67571244

INTERVENTIONS:
Drug: JNJ-67571244 — JNJ-67571244 will be administered.

SUMMARY:
The main purpose of this study are to determine the recommended Phase 2 dose(s) (RP2D) route of administration, schedule and the maximum tolerated dose (MTD) in Part 1 and to determine the safety and tolerability of JNJ-67571244 at the RP2D regimen(s) and to evaluate the preliminary clinical activity of JNJ-67571244 in Part 2.

DETAILED DESCRIPTION:
This is first-in-human (FIH) Phase 1, open-label, multicenter, dose escalation study with dose expansion to evaluate the safety, tolerability, and preliminary antitumor activity of JNJ-67571244 in adult participants with relapsed or refractory acute myeloid leukemia (AML) or high-risk or very high-risk myelodysplastic syndromes (MDS) who are ineligible for or have exhausted standard therapeutic options. The study is divided into 3 periods: a Screening Phase (within 28 days before the first dose of study drug), a Treatment Phase (first dose of study drug until the last dose of study drug) and a Post-treatment Follow-up Phase (up to the end of study participation or end of study). Duration of study is 2.3 years.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of:

  a) Acute Myeloid Leukemia (AML) according to the World Health Organization 2008 criteria with relapsed or refractory disease and ineligible for or have exhausted standard therapeutic options b) high-risk or very high-risk Myelodysplastic Syndrome (MDS) according to International Prognostic Scoring System (IPSS-R) and relapsed or refractory after at least 1 course of hypomethylating therapy and ineligible for or have exhausted standard therapeutic options per investigator discretion should be included
* Eastern Cooperative Oncology Group (ECOG) performance status grade of 0 or 1
* Women of childbearing potential must have a negative pregnancy test at screening and prior to the first dose of study drug using a highly sensitive pregnancy test (either serum or urine beta human chorionic gonadotropin [beta-hCG])
* Chemistry laboratory parameters within the following range during screening:

  a) aspartate transaminase (AST) and alanine aminotransferase (ALT) less than or equal to (<=) 3* upper limit of normal (ULN), b) Total bilirubin <=1.5*ULN; participants with congenital bilirubinemia, such as Gilbert's syndrome, may enroll if conjugated bilirubin is within normal range, c) Creatinine clearance calculated or measured creatinine clearance greater than or equal to (>=) 30 milliliters per minute (mL/min)
* Before the first dose of study drug:

  1. Women of childbearing potential and fertile men who are sexually active must agree to use a highly effective method of contraception (less than [<] 1 percent {%} year failure rate from the time of signing the informed consent form [ICF]) during the study and for 90 days after the last dose of study drug. Contraception must be consistent with local regulations regarding the use of birth control methods for participants participating in clinical trials. 1) Participant must agree to practice a highly effective method of contraception (failure rate of <1% per year when used consistently and correctly). Examples of highly effective contraceptives include: a) user-independent methods: implantable progestogen-only hormone contraception associated with inhibition of ovulation; intrauterine device; intrauterine hormone-releasing system; vasectomized partner; b) user-dependent methods: combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, and transdermal; progestogen-only hormone contraception associated with inhibition of ovulation: oral and injectable, c) In addition to the highly effective method of contraception, a man: 1) Who is sexually active with a woman of childbearing potential must agree to use a barrier method of contraception (for example, condom with spermicidal foam/gel/film/cream/suppository), 2) Who is sexually active with a woman who is pregnant must use a condom, c) Women and men must agree not to donate eggs (ova, oocytes) or sperm, respectively, during the study and for 90 days after the last dose of study drug

Exclusion Criteria:

* Willing and able to undergo allogenic stem cell transplant <=6 months before the first dose of study drug, has evidence of graft versus host disease, or requires immunosuppressant therapy (exception: daily doses less than 10 milligram (mg) prednisone or equivalent are allowed for adrenal replacement)
* For Part 1 only, prior treatment with CD33 targeting therapy targeting T-cell redirection (for example, CD-3 redirection technology or chimeric antigen receptor [CAR]-T-cell therapy)
* For Part 1 only, prior Grade 3 cytokine release syndrome (CRS) related to any T-cell redirection (for example, CD-3 redirection technology or CAR-T cell therapy)
* Prior treatment with a checkpoint inhibitor such that the first dose of JNJ-67571244 would occur within less than 5 half-lives. Prior treatment with chemotherapy, targeted therapy, immunotherapy, radiotherapy, or treatment with an investigational anticancer agent, an investigational drug (including investigational vaccines), within 2 weeks prior to the first dose or at least 4 half-lives, whichever is less, or currently receiving investigational therapy in a clinical trial. Hydroxyurea may be used
* Toxicities (except for alopecia, peripheral neuropathy, thrombocytopenia) from previous anticancer therapies that have not resolved to baseline levels or to Grade 1 or less

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2022-03-26 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Part 1 and Part 2: Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 100 days after the last dose of study drug or until the start of a subsequent anticancer therapy, whichever comes first (that is up to 2.3 years)
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Part 1: Number of Participants with Dose-Limiting Toxicity (DLTs) | Up to 28 days
  Number of participants with dose-limiting toxicity will be assessed. The DLTs are based on drug-related adverse events and defined as any of the following events: infusion-related reactions, non-hematologic toxicity of Grade 3 or higher, or hematologic toxicity.
Part 1: Severity of DLT as Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) | Up to 28 days
  The DLT evaluation period is defined as the first 28 days after a participant's first infusion (Day 1). Severity criteria is based on Grade 1, 2, 3, 4 and 5, will be assessed by the investigator as per below grades. Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening consequences; Grade 5: Death related to adverse event.
Part 2: Overall Response Rate (ORR) | Approximately 2.3 years
  ORR is defined as the percentage of participants who have complete response (CR) and incomplete blood count recovery (CRi) (AML) or CR and partial response (PR) (MDS) as per modified International Working Group response (IWGR) criteria.

SECONDARY OUTCOMES:
Part 1 and Part 2: Serum Concentrations of JNJ-67571244 | Approximately 2.3 years
  Serum samples will be analyzed to determine concentrations of JNJ-67571244 using a validated immunoassay method.
Part 1 and 2: Systemic Cytokine Concentrations | Approximately 2.3 years
  Serum cytokine (Interleukin [IL]-2, IL-6, IL-8, IL-10, and Interferon [IFN]-alpha, IFN-delta with same unit of measurement) concentrations will be measured for biomarker assessment.
Number of Participants with Depletion of CD33-Expressing Cells | Approximately 2.3 years
  Number of participants with depletion of CD33-expressing cells will be assessed.
Part 1 and 2: Concentration of Markers of T-Cell Activation | Up to 24 days
  Levels of T-cell activation marker CD25 will be reported as measured by flow cytometry and cytometry by time of flight (CyTOF). T-cell activation will also be assessed by measuring cytokine release.
Part 1 and 2: Number of Participants with JNJ-67571244 Antibodies | Week 1 (Day 1) up to post treatment Week 8
  Anti-JNJ-67571244 antibodies will be evaluated in serum samples collected from all participants and the titer of confirmed positive samples will be reported.
Part 1 and Part 2: Duration of response (DOR) | Approximately 2.3 years
  DOR is calculated from date of initial documentation of a response (complete response (CR) and incomplete blood count recovery (CRi) (AML) or CR and partial response (PR) [MDS]) to the date of first documented evidence of relapse, defined in disease-specific response criteria, or death, whichever occurs first.
Part 1 and Part 2: Time to response (TTR) | Approximately 2.3 years
  TTR defined for the responders as the time from the date of first dose of study drug to the date of initial documentation of a response (CR and CRi [AML] or CR and PR [MDS]), as defined in the disease-specific response criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (17):
- United States (9):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - NYU Hematology Associates, New York, New York
  - Levine Cancer Institute, Carolinas HealthCare System, Charlotte, North Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Germany (3):
  - Universitaetsklinikum Leipzig, Leipzig
  - Klinikum der Universitaet Muenchen, München
  - Universitätsklinikum Münster; Med. Klinik A - Germany, Münster
- Spain (5):
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp. Virgen Del Rocio, Seville

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency